CLINICAL TRIAL: NCT01290003
Title: Role of Prophylactic Antibiotics in Preventing Neonatal Sepsis in Neonates Born Through Meconium Stained Amniotic Fluid - A Randomized Controlled Trial
Brief Title: Role of Antibiotics in Preventing Infection in Babies Born Through Meconium Stained Liquor
Acronym: AbProM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lady Hardinge Medical College (Other Government)
Responsible Party: Principal Investigator, Sushma Nangia, M.D., Professor Pediatrics, Lady Hardinge Medical College
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: LHMC/054/Ab-Pro-M
Record Dates: First submitted 2011-02-03; First posted 2011-02-04 (Estimated); Last update posted 2015-09-29 (Estimated); Status verified 2015-09

CONDITIONS: Neonatal Sepsis
Keywords: Antibacterial agents; Neonate; Meconium stained amniotic fluid; Neonatal sepsis
MeSH Terms: conditions — Neonatal Sepsis | interventions — Piperacillin, Tazobactam Drug Combination; Amikacin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Antibiotic Group (Experimental): Neonates randomized to intervention Group(Antibiotic group)will receive the first line antibiotics (Piperacillin-Tazobactam and Amikacin) as per the unit policy for 72 hours. These neonates will also be monitored by performing sepsis screens and blood culture for development of sepsis.
  Interventions: Drug: Piperacillin-Tazobactam and Amikacin
- No Antibiotic Group (No Intervention): Neonates randomized to 'No antibiotic group' will receive supportive treatment as per standard unit protocol. These neonates will be monitored by performing sepsis screens and blood culture for development of sepsis.

INTERVENTIONS:
Drug: Piperacillin-Tazobactam and Amikacin — Inj Piperacillin-Tazobactam 50 mg/Kg/dose 12 hourly IV X 3 days (6 doses) Inj Amikacin 15 mg/kg/dose 24 hourly IV X 3 days (3 doses)
  Arms: Antibiotic Group

SUMMARY:
The purpose of the study is to evaluate the role of antibiotics in preventing infection in babies born through meconium stained amniotic fluid. Normally babies do not pass meconium while in utero. In response to hypoxic stress babies may pass meconium before birth and are likely to be candidates for problems related to meconium passage and its inhalation. It is believed that these babies are more prone to infections as meconium enhances bacterial growth and may predispose such babies to secondary bacterial infections. In addition, meconium passage has been incriminated as a pointer of in-utero infection. Whether use of antibiotics in babies born through meconium stained amniotic fluid will reduce the infectious episodes and complications thereof or not is not clear. Moreover, there is not much published literature to prove or refute the same. Most clinicians have a low threshold for using antibiotics in such babies. In view of the uncertainty regarding antibiotic usage in these babies, the investigators decided to investigate the role of prophylactic antibiotics in prevention of neonatal sepsis in babies born through meconium stained amniotic fluid.

DETAILED DESCRIPTION:
Meconium passage in newborn infants is a developmentally programmed event normally occurring within first 24-48 hours of birth. Intra uterine meconium passage in near term or term fetuses has been associated with feto-maternal stress factors and/or infections, whereas meconium passage in post term pregnancies has been attributed to gastro-intestinal maturity. The meconium staining of amniotic fluid occurs in 12% of all live births per annuum. Aspiration of meconium that occurs during intra uterine life or after delivery with the first few breaths may result in or contribute to respiratory pathology known as meconium aspiration syndrome (MAS) which represents a leading cause of the perinatal morbidity, occurring in 5-20% of all babies born through MSAF.

The routine use of antibiotics in MSAF babies has been advocated for a long time as a part of the conventional treatment. Meconium passage in utero is hypothesized to represent a response to fetal bacterial infection in addition to intrauterine hypoxia. Additionally the rationale for use of antibiotics includes the radiographic similarity of MAS to bacterial pneumonia, in vitro enhancement of bacterial growth in presence of meconium as well as the possibility of meconium induced inhibition of phagocytic activity and respiratory burst response by alveolar macrophages rendering patients with MAS more susceptible to infection. These recommendations however are empirical and the incidence of bacterial infection in neonates born through MSAF as well as in MAS has not been systematically evaluated, to date. With the rising concern about the emergence of resistant strains in neonatal ICUs and the possible side effects of antibiotics (like amino glycosides) including nephrotoxicity and ototoxicity in neonates, a systematically conducted, randomized controlled trial is necessary to assess the utility of antibiotics in the routine management of infants with MSAF and MAS. Hence the purpose of this prospective randomized controlled trial is to compare the clinical course, complications, and infection related outcomes in cases of MSAF and MAS, treated with or without antibiotics therapy

ELIGIBILITY:
Inclusion Criteria:

* Gestation > 37 weeks
* Meconium staining of amniotic fluid
* Cephalic presentation
* Singleton pregnancy

Exclusion Criteria:

* Major Congenital malformation
* Refusal of consent

Ages: 30 Minutes to 2 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 250 (Actual)
Dates: Start 2010-06; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Incidence of sepsis | First 28 days of life
  Incidence of sepsis in first 28 days defined as -
  1. SUSPECTED SEPSIS - Sepsis Screen > 2 parameters positive and/or
  2. CONFIRMED SEPSIS - Sepsis Screen positive + Blood or CSF culture positive for bacteria.
  Sepsis Screen
  1. Total leukocyte count < 5000/mm3
  2. Absolute neutrophil count < 1800/cu.mm.(Low counts as per Monroe chart for term neonates)
  3. Immature/total neutrophil ratio > 0.2
  4. Micro-ESR > 15mm in 1st hour
  5. C Reactive Protein (CRP) > 1 mg/dl

SECONDARY OUTCOMES:
Mortality; | First 28 days of life
Respiratory support; | Till discharge from the hospital
  1. Requirement of respiratory support
  2. The mode of respiratory support viz. Supplemetal Oxygen therapy, CPAP, Mechanical ventilation, High Frequency ventilation
  3. Duration of each kind of respiratory support required
Duration of Hospital stay | Till discharge
Complications | Till discharge
  Incidence of PPHN by Echocardiography, Pneumothorax by transillumination confirmed by chest x-ray, azotemia by Kidney function test panel

CONTACTS AND LOCATIONS:
Overall Officials: Sushma Nangia, MBBS, MD, DM, Study Chair — Lady Hardinge Medical College, New Delhi, India
Locations (1):
- Kalawati Saran children's Hospital, Lady Hardinge Medical College, New Delhi, National Capital Territory of Delhi, India

REFERENCES:
- [Derived] Goel A, Nangia S, Saili A, Garg A, Sharma S, Randhawa VS. Role of prophylactic antibiotics in neonates born through meconium-stained amniotic fluid (MSAF)--a randomized controlled trial. Eur J Pediatr. 2015 Feb;174(2):237-43. doi: 10.1007/s00431-014-2385-4. Epub 2014 Aug 3. PMID 25084971